CLINICAL TRIAL: NCT04422262
Title: Impact of the Italian Lockdown on Lifestyles and Psychosocial Status of the Moli-Sani Study Cohort and the Italian General Population
Brief Title: Analysis of Long Term Risk of Coronavirus Disease-19 Emergency
Acronym: ALTRISCOVID-19
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: DEP 1/2020
Record Dates: First submitted 2020-05-24; First posted 2020-06-09 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Lifestyle; Dietary Habits; Psychosocial Problem
Keywords: pandemic; lockdown; lifestyles; dietary habits; psychosocial factors
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Moli-sani Study sub-cohort: A sample of 2,500 men and women from the Moli-sani Study cohort (2005-2010) who were re-examined in 2017-2020. Participants will be contacted by telephone by researchers of the Moli-sani Study recruitment team in order to collect dietary, lifestyle and psychosocial information and assess potential changes possibly occurred during Phase 1 lockdown.
- Italian general population: The project will retrospectively collect data through a web-based survey using Google form. The questionnaire consists of the same items used for the Moli-sani sub-cohort. The project aims at including as many subjects' records as possible.

SUMMARY:
The aim of this study is to investigate dietary, lifestyle and psychosocial changes possibly occurred during Italy's lockdown, that is in the period of time between March 9 2020 and May 3 2020 (hereafter referred to as the Phase 1 lockdown) in two different populations: the Moli-sani Study cohort and the Italian general population.

DETAILED DESCRIPTION:
The containment measures released by the Italian Government for the period between March 9- May 3 2020 have been aimed to reduce the movement of people from their homes, which was only allowed in cases of special need, and the use of smart work (working from home) wherever possible .As a consequence, the lockdown period is likely to have lasting effects on people and their lifestyles, especially nutrition, and psychosocial well-being.

A web-based questionnaire was developed to retrospectively investigate dietary, lifestyle and psychosocial changes possibly occurred during Italy's lockdown, that is in the period of time between March 9 2020 and May 3 2020 (hereafter referred to as the Phase 1 lockdown).

The potential impact of Phase 1 lockdown on lifestyles will be tested in two distinct population cohorts, that is the Moli-sani Study cohort (established among residents in the Molise region in the period 2005-2010) and a sample of the general Italian population, aged ≥ 18 years.

ELIGIBILITY:
Inclusion Criteria for the Moli-sani Study sub-cohort:

* Re-examination in 2017-2020;
* Able to give verbal consent

Exclusion criteria for the Moli-sani Study sub-cohort:

- Not able to give verbal consent

Inclusion Criteria for the General Italian population cohort:

* Age >= 18 years.
* All subjects from the general population with access to electronic devices and the Internet (e.g. personal computer, smartphone) and is fluent in Italian will be eligible.

Exclusion Criteria for the General Italian population cohort:

* Subjects younger than 18 years
* Only people with access to personal computers, smartphones and the Internet, and fluency in Italian will be able to participate. These exclusions are not based on age, gender, pregnancy, racial, or ethnic origin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moli-sani Study sub-cohort A sample of 2,500 men and women from the Moli-sani Study cohort (2005-2010) who were re-examined in 2017-2020. Participants will be contacted by telephone by researchers of the Moli-sani Study recruitment team in order to collect dietary, lifestyle and psychosocial information and assess potential changes possibly occurred during Phase 1 lockdown. This project will be hereafter referred to as Moli-LOCK Study.
  Italian general population The project will retrospectively collect data through a web-based survey using Google form. The questionnaire consists of the same items used in the Moli-LOCK Study. The investigators aim at including as many subjects' records as possible. This project will be hereafter referred to as ALT RISCOVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 4307 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessing changes in smoking status during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential modifications in smoking habits, by administering specific questions on how and to what extent this behavior has been modified during lockdown.
  The questions will investigate whether during the Italian lockdown smokers have increased the daily number of cigarettes, or whether they quitted, and whether nonsmokers have started to smoke and to what extent.
Assessing changes in physical activity during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential modifications in physical activity, by administering specific questions on how and to what extent this behavior has been modified during lockdown.
  The questions will investigate whether during the Italian lockdown subjects have experienced a reduction of their usual exercise in terms of minutes per week.
Assessing changes in work-related activities during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential modifications in working and work-related activities, by administering specific questions on how and to what extent work-related issues have been modified during lockdown.
  The questions will investigate whether during the Italian lockdown subjects have shifted to smart working, experienced job loss/reduction, salary reductions, used public transport to go to work.
Assessing changes in social habits during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential modifications in social life, by administering specific questions on how and to what extent social habits have been modified during lockdown.
  The questions will investigate how often during the Italian lockdown subjects used to go out on average during the week, and on what occasions they were used to use masks.

SECONDARY OUTCOMES:
Assessing changes in dietary habits during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential modifications in frequency consumption of several food groups, with a specific focus on those typical of a Mediterranean diet, by administering specific questions on whether the consumption of several food groups have been modified during lockdown. The questions are 'Please indicate whether the consumption of each of the following foods has been changed during the lockdown as compared to your usual intake'. Possible answers are 'not changed', 'increased' or 'decreased'.
Assessing depression during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential development of depressive symptoms during the Italian lockdown by administering the Patient Health Questionnaire- 9 (PHQ-9) .
Assessing anxiety during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential onset of anxiety during the Italian lockdown by administering the Generalized Anxiety Disorder scale (GAD-7).
Assessing stress during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential onset of stress during the Italian lockdown by administering the Perceived stress scale (PSS-4).
Assessing post-traumatic stress disorder during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate potential onset of post-traumatic stress disorder during the Italian lockdown by administering the Screening Questionnaire for Disaster Mental Health -SQD.
Assessing social support during Italian lockdown | From March 9 2020 to May 3 2020
  The study will evaluate social support through questions asking how much during the lockdown period people could count on the support / help of people (e.g. relatives, friends, neighbors, health care professionals, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: No